CLINICAL TRIAL: NCT00691067
Title: A Randomized, Double-blind Placebo-controlled Crossover Trial of Mifepristone in Gulf War Veterans With Chronic Multisymptom Illness
Brief Title: A Controlled Trial of Mifepristone in Gulf War Veterans With Chronic Multisymptom Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bronx Veterans Medical Research Foundation, Inc (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julia Golier, Clinical Director, Mental Health Patient Care Center, Bronx Veterans Medical Research Foundation, Inc
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GW060048
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Multisymptom Illness in Gulf War Veterans
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone (Experimental): 600mg of Mifepristone
  Interventions: Drug: mifepristone
- Placebos (Placebo Comparator): Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: mifepristone — 200 mg po per day x 6 weeks
  Arms: Mifepristone
Drug: Placebos — placebo
  Arms: Placebos

SUMMARY:
We propose to conduct placebo-controlled trial of the glucocorticoid receptor antagonist mifepristone in Gulf War veterans (GWV) with chronic multisymptom illness (CMI) to examine its effects on physical and mental health and cognitive functioning. In addition, we propose to examine whether HPA axis biomarkers or their response to mifepristone are useful predictors of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the 1991 Gulf War
* Veteran meets criteria for multisymptom illness

Exclusion Criteria:

* Veteran lacks the capacity to provide consent.
* Veteran has a major medical or neurological disorder or traumatic brain injury
* Veteran has morning plasma cortisol level less than 5 mcg/dl or a history of adrenal insufficiency
* Veteran is taking oral corticosteroids
* Veteran has a lifetime diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder
* Veteran has been psychiatrically hospitalized or attempted suicide within the previous 2 years
* Veteran has current suicidal ideation
* Veteran is pregnant or breastfeeding or plans to become pregnant within the year (male or female) not willing to use appropriate forms of contraception during the study and for at least 90 days post treatment.
* Women veterans with diseases of the uterus by history or a family history of uterine cancer
* Known allergy to mifepristone

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
change in the health components score of the veterans RAND 36-item health survey (VR-36) | baseline, every two weeks, endpoint

SECONDARY OUTCOMES:
cognitive functioning and measures of depression, fatigue and PTSD | baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Golier, M.D., Principal Investigator — James J Peters VA Medical Center
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Golier JA, Caramanica K, Michaelides AC, Makotkine I, Schmeidler J, Harvey PD, Yehuda R. A randomized, double-blind, placebo-controlled, crossover trial of mifepristone in Gulf War veterans with chronic multisymptom illness. Psychoneuroendocrinology. 2016 Feb;64:22-30. doi: 10.1016/j.psyneuen.2015.11.001. Epub 2015 Nov 10. PMID 26600007